CLINICAL TRIAL: NCT01546441
Title: IMPACT Plus: The Integrated Complex Care Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Aging
Keywords: primary care; aging; interprofessional care; multimorbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interprofessional assessment (Experimental): patients receive an interprofessional assessment in a team environment
  Interventions: Behavioral: interprofessional assessment
- usual care (Active Comparator): Usual care in family practice
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: interprofessional assessment — assessment by interprofessional team
  Arms: interprofessional assessment
Behavioral: usual care — usual care in primary care clinic
  Arms: usual care

SUMMARY:
The "IMPACT Plus" Integrated Complex Care Clinic will create a team model of simultaneous interprofessional consultation and planning that brings together patients with complex or multiple chronic diseases, significant others/caregivers, the primary care team, community care providers and, uniquely, secondary consultation in real time at the primary care site. The purpose of this study is to evaluate whether the IMPACT clinic will reduce admission to hospital and visits to the emergency department (ED) in comparison to a control (usual care) group during a one year period of observation. Chart audits will be conducted on a monthly basis to calculate patients' complexity scores and data on all health services provided during the intervention phase, and compared between the intervention and control group. Additionally, surveys and semi-structured interviews aimed to measure patient, caregiver, and healthcare professional satisfaction of the IMPACT+ prior to and after initial assessment will be collected.

DETAILED DESCRIPTION:
The investigators propose a pragmatic clinical trial to evaluate whether the IMPACT model will reduce hospital admissions and emergency room visits. All patients who meet the eligibility criteria will be randomized to be invited for assessment in IMPACT or be followed in usual care. Each FHT will generate a list of eligible participants drawn from their EMR. Participants will be randomly selected from this list and patients will be invited for an IMPACT assessment. Using data collected at each FHT by a trained chart abstractor on a monthly basis, all hospital admissions and emergency room visits will be counted. As well, all health service utilization for both intervention and control group will be collected. The investigators will compare the proportion of patients admitted to hospital or seen in the emergency room between the intervention and control group for the one year time period. For the secondary objectives of the study, patient and care givers in the intervention group will be asked to complete the Caregiver Strain Index (a standardized and validated instrument) both before the IMPACT intervention and up to 6 months later. The investigators will adapt an existing survey to measure health care professionals' experiences in providing care in an inter-professional team for seniors with complex chronic illness. The Dimensions of Teamwork Survey, will be administered at each FHT at the beginning of the study and at the end of the intervention period in order to assess team function and stability of team function. Lastly, interviews with patients, caregivers, and healthcare professionals will be conducted to explore satisfaction with the IMPACT experience and subsequent care as well as self-efficacy in managing their care. The interviews will be audio-recorded and professionally transcribed. Key themes emerging from the qualitative data will be identified. Preliminary findings will be subjected to a process of member checking/respondent validation to ensure accuracy of interpretation.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are as follows:

  * 65 years of age or older;
  * three or more chronic diseases requiring monitoring and treatment (or two chronic diseases when one is frequently unstable);
  * five or more long-term medications;
  * a minimum of one ADL limitation; and
  * approval by family physician as suitable for IMPACT assessment.

Exclusion Criteria:

* The exclusion criteria are as follows:

  * previous IMPACT assessment; or
  * deemed not suitable by family physician.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Hospital Admissions | 6 months
  We will compare the hospitalization rates between those who have received and those who have not received the intervention

SECONDARY OUTCOMES:
Emergency room visits | 6 months
  we will compare the rate of emergency room visits between those who received and those who did not receive the intervention